## **Study Title:**

Cognitive Enhancement through Transcranial Laser Therapy (LLLT)

Clinicaltrials.gov Registration Number: NCT02851173

**Date of Document:** 10/15/2014

## 1. Title:

Cognitive Enhancement through Transcranial Laser Therapy

## 2. Principal Investigator:

Name: Andreana Haley

EID: aph355

Department: Psychology

## **Statistical Plan:**

- 1. Primary outcome measure (PVT) will be analyzed using mixed ANOVA with 1 between-subjects factor (Treatment Group) and 1 within subjects factor (Time). Cognitively unimpaired (CU) and MCI groups will be analyzed separately. The contrast of interest will be Treatment Group by Time interaction. Alpha level of significance will be set at 0.05.
  - a. Secondary outcome measures (2Back performance, % Correct and Reaction Time) will be analyzed using mixed ANOVA with 1 between-subjects factor (Treatment Group) and 1 within subjects factor (Time). Cognitively unimpaired (CU) and MCI groups will be analyzed separately. The contrast of interest will be Treatment Group by Time interaction. Alpha level of significance will be set at 0.05.
  - b. Secondary outcome measures (2Back activation intensity within 8 *a priory* ROIs) will be analyzed using mixed ANOVA with 1 between-subjects factor (Treatment Group) and 1 within subjects factor (Time), only for participants who can perform the task to criterion (%Correct>50%). Cognitively unimpaired (CU) and MCI groups will be analyzed separately. The contrast of interest will be Treatment Group by Time interaction. Alpha level of significance will be set at 0.05 due to the exploratory nature of the analysis.
  - c. A priori ROIs were chosen based on prior literature. They are as follows:

| ROI# | x | y | z | size (mm2) | designation |
|---|---|---|---|---|---|
| 1 | -33 | 4 | 56 | 2087 | Left middle frontal gyrus |
| 2 | -5 | 19 | 44 | 1651 | Left medial frontal/superior frontal gyrus |
| 3 | 37 | -63 | 53 | 683 | Right superior parietal lobule |
| 4 | -49 | -52 | 44 | 1333 | Left inferior parietal lobule |
| 5 | -44 | 45 | 13 | 1139 | Left middle frontal gyrus |
| 6 | 33 | 48 | 15 | 955 | Right superior frontal gyrus |
| 7 | 32 | 5 | 55 | 553 | Right middle frontal gyrus |
| 8 | 47 | 14 | 3 | 335 | Right inferior frontal gyrus |